CLINICAL TRIAL: NCT05242146
Title: A Phase 1b/2, Open-label Dose Escalation With Expansion Study of GB5121 in Adult Patients With Relapsed/Refractory Primary or Secondary Central Nervous System Lymphoma or Primary Vitreoretinal Lymphoma, With a Phase 2 Open-label Single Dose Level Study of GB5121 in Adult Patients With Relapsed/ Refractory Primary Central Nervous System Lymphoma
Brief Title: GB5121 in Adult Patients With Relapsed/Refractory CNS Lymphoma
Acronym: STAR CNS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: GB005, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB5121-2101
Record Dates: First submitted 2022-01-31; First posted 2022-02-16 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: CNS Lymphoma
Keywords: R/R PCNSL; SCNSL; PVRL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GB5121 (Experimental): GB5121 orally twice per day (BID)
  Interventions: Drug: GB5121

INTERVENTIONS:
Drug: GB5121 — Capsule containing GB5121

SUMMARY:
The STAR CNS trial is a 3-part study, comprising a phase 1b dose escalation, dose expansion, and a phase 2, to assess the safety, tolerability, dose-limiting toxicity(ies), maximum tolerated dose, and/or optimal biological dose, determine the recommended phase 2 dose, preliminary anti-tumor activity and efficacy of the recommended phase 2 dose of GB5121.

DETAILED DESCRIPTION:
Note: The Phase 1b dose expansion and Phase 2 parts of the study were not initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically/cytologically confirmed primary central nervous system lymphoma (PCNSL), primary vitreoretinal lymphoma (PVRL), or CNS-only involvement of a systemic B-cell lymphoma.
2. All patients must have relapsed/refractory disease and must have received all possible standard-of-care CNS-directed therapy treatment regimens or patients for which further standard-of-care treatment options are contraindicated or declined.
3. Patients must be able to tolerate gadolinium-enhanced magnetic resonance imaging (MRI) scans, or contrast-enhanced computed tomography (CT).
4. Patients with parenchymal lesions must have baseline imaging (gadolinium-enhanced MRI or if contraindicated, contrast-enhanced CT, of the brain) within 28 days prior to first study drug dose. For patients with leptomeningeal disease only, cerebrospinal fluid (CSF) cytology must document lymphoma cells and/or imaging findings consistent with leptomeningeal disease after informed consent and prior to first study dose (at the discretion of the Investigator).
5. Patients with parenchymal lesions must have measurable disease (disease that has at least one lesion on imaging ≥ 10 mm in the longest diameter) on imaging (gadolinium-enhanced MRI or if contraindicated, contrast-enhanced CT, of the brain) prior to first study dose.
6. Patients must be able to tolerate and consent for a lumbar puncture and/or have pre-existing placement of an Ommaya reservoir, unless clinically contraindicated.
7. Patients must have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Demonstrate adequate bone marrow and organ function.

Exclusion Criteria:

1. Patients are concurrently using other approved or investigational antineoplastic agents.
2. Patients have an active concurrent malignancy requiring active therapy.
3. Patients are allergic to components of the study drug.
4. Patients have a known bleeding diathesis (eg, von Willebrand's disease) or hemophilia.
5. Patients who require therapeutic anticoagulation, including dual antiplatelet agents. Patients who have received therapeutic anticoagulation, including dual antiplatelet agents, within 5 half-lives of the anticoagulant or 14 days, whichever is longer, prior to starting the study drug. Patients who require the use of antiplatelet agents should be discussed with the Sponsor's Medical Monitor.
6. Patients have significant abnormalities on screening electrocardiogram (ECG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, uncontrolled hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening.
7. Patients with any of the following will be excluded:

   1. A marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval > 480 ms [CTCAE grade 2]) using Frederica's QT correction formula.
   2. A history of additional risk factors for Torsades de Pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
   3. The use of concomitant medications that prolong the QT/QTc interval.
8. Patients are known to have a history of active or chronic infection with hepatitis C virus (HCV), hepatitis B virus (HBV), as determined by serologic tests.
9. Known history of infection with human immunodeficiency virus (HIV).
10. Patients are known to have an uncontrolled active infection.
11. Patients have a history of stroke or intracranial hemorrhage within 6 months prior to enrollment.
12. Patients have a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the Investigator, could compromise the subject's safety or put the study outcomes at undue risk.
13. Women who are pregnant or nursing (lactating).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Phase 1b Dose Escalation - Incidence of Adverse Events | From first dose until 28 days after the last dose of GB5121
Phase 1b Dose Escalation - Dose Limiting Toxicity(ies) | From Cycle 1, Day 1 through Cycle 1, Day 28 inclusive, Each Cycle=28 days
Phase 1b Dose Escalation - Serious Adverse Events | From consent until 28 days after the last dose of GB5121
Phase 1b Dose Escalation - Optimal Biologic Dose and/or Maximum Tolerated Dose and Recommended Phase 2 Dose | From first dose up to approximately 36 months
Phase 1b Dose Expansion - Incidence of Adverse Events | From first dose until 28 days after the last dose of GB5121
Phase 1b Dose Expansion - Serious Adverse Events | From consent until 28 days after the last dose of GB5121
Phase 2 - Objective Response Rate According to International Primary CNS Lymphoma Collaborative Group (IPCG) Criteria by Blinded Independent Central Review Committee (BICR) | From Study Day 1 until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months

SECONDARY OUTCOMES:
Phase 1b Dose Expansion - Objective Response Rate According to IPCG Criteria by Investigator Assessment | From Study Day 1 until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Duration of Response by BICR Committee | From first observation of complete response, unconfirmed complete response or partial response until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Confirmed Complete Response by BICR Committee | From Study Day 1 until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Objective Response Rate According to the IPCG Criteria by Investigator Assessment | From Study Day 1 until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Median Progression-Free Survival | From Study Day 1 until disease progression assessed by the Investigator per IPCG criteria, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Progression-Free Survival at Week 24 | From Study Day 1 until Week 24
Phase 2 - Median Overall Survival | From Study Day 1 until death, unacceptable toxicity, or discontinuation, up to approximately 36 months
Phase 2 - Incidence of Adverse Events | From first dose until 28 days after the last dose of GB5121
Phase 2 - Incidence of Serious Adverse Events | From consent until 28 days after the last dose of GB5121

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center Main Campus, New York, New York
- Australia (2):
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- The Ottawa Hospital, Ottawa, Ontario, Canada
- France (5):
  - South Lyon Hospital Center, Pierre-Bénite, Lyon
  - Bergonie Institute, Bordeaux, Nouvelle-Aquitaine
  - CHU APHM la Timone / Aix Marseille University, Marseille, Provence-Alpes-Cote d'Azure
  - La Pitie-Salpetriere University Hospital, Paris, Île-de-France Region
  - Institut Curie Site Saint-Cloud, Saint-Cloud, Île-de-France Region
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Middlemore Hospital, Papatoetoe, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No